CLINICAL TRIAL: NCT05191810
Title: Efficacy of Educational Intervention as Supporting Element in the Treatment of Functional Constipation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Dziechciarz, MD, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZAPWUM11/2021
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Constipation - Functional
Keywords: fluid intake; functional constipation; children; PEG; macrogol; educational intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Macrogol (PEG 3350, PEG 4000), standard dosage Educational intervention: Recommendation of adequate for age fluid intake plus standard information about non-pharmacological supporting treatment
  Interventions: Behavioral: Educational information
- Control Group (No Intervention): Macrogol (PEG 3350, PEG 4000), standard dosage Standard educational information about non-pharmacological supporting treatment

INTERVENTIONS:
Behavioral: Educational information — Educational information about non-pharmacological supporting treatment of functional constipation, involving recommendation of adequate for age fluid intake
  Arms: Study Group

SUMMARY:
The purpose of this study is to determine whether educational intervention (recommendation of adequate fluid intake) is effective as an element supporting the treatment of functional constipation in children.

DETAILED DESCRIPTION:
Constipation is a common condition in children which affects around 10% of the paediatric population. In 95 % cases it is a functional disorder of the digestive tract, without any organic cause. Recommendations of lifestyle modifications accompanying pharmacological treatment of constipation are very popular among healthcare providers, although there is limited data concerning non-pharmacological treatment methods of this condition. Adequate for age fluid intake is now recommended for patients with constipation. Further research is needed to form stronger recommendations in the future. The purpose of this study is to determine whether educational intervention (recommendation of adequate fluid intake) is effective as an element supporting the treatment of functional constipation in children.

ELIGIBILITY:
Inclusion Criteria:

Children with functional constipation diagnosed based on Rome IV criteria

Exclusion Criteria:

1. Children with organic causes of constipation; eg, anorectal malformations, or Hirschsprung's disease
2. Children who fulfil the criteria of Irritable Bowel Syndrome
3. Significant, unstabilised chronic health conditions requiring major drug adjustment during the last 3 months.
4. Unintentional weight loss greater than or equal to 5% of their body weight within the last 3 months
5. Recurrent or unexplained fevers
6. History of abdominal surgery involving the luminal gastrointestinal tract, except appendectomy, or hernia repairs
7. Concomitant use of drugs that are known to affect gastrointestinal motility
8. Established diagnoses of autism spectrum disorders
9. Mental retardation
10. Children who are exclusively breastfed
11. Non-retentive faecal incontinence

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-07 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who no longer fulfill the Rome IV constipation criteria | last week of intervention
  Success of therapy defined as no longer fulfilling the Rome IV constipation criteria during the last week of intervention.

SECONDARY OUTCOMES:
Average daily fluid intake (ml) before the beginning of the intervention and during the last week of intervention | 8 weeks
  Assessed by a 2-day food and fluid intake diary made by patient and/or caregiver at the beginning of the intervention and during the last week of intervention
Frequency (number per week) of bowel movements during the fourth and last weeks of intervention | 8 weeks
  One of the Rome IV constipation criteria
Frequency of fecal incontinence (number per week) during the fourth and last weeks of intervention | 8 weeks
  One of the Rome IV constipation criteria
Painful bowel movements (number per week) during the fourth and last weeks of intervention | 8 weeks
  One of the Rome IV constipation criteria
Stomachache and bloating (number of episodes per week) during the fourth and last weeks of intervention | 8 weeks
  Symptoms related to constipation
Macrogol dose (mg/kg/day) during the fourth and last weeks of intervention | 8 weeks
  Macrogol dose needed to achieve treatment success (no longer fulfilling the Rome IV constipation criteria).
Need for rescue laxative treatment during the intervention (number of cases) | 8 weeks
  In case of lack of bowel movements for three consecutive days, the macrogol dose will be augmented to 1-1.5g/kg/day until a bowel movement occurs.
Time (days) from the start of intervention needed to achieve treatment success. | 8 weeks
  Time needed to no longer fulfill the Rome IV constipation criteria
Adverse events during intervention (number and type of reported adverse events) | 8 weeks
  Any adverse events reported by the patient or caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Dziechciarz, MD PhD, Principal Investigator — Department of Pediatrics of the Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data on request via e-mail
Supporting Information: Study Protocol, ICF
Time Frame: 1.01.2022-31.12.2024
Access Criteria: we plan to share all individual patients data on every outcome measure on request from any other researcher after completion of the study

REFERENCES:
- [Background] Koppen IJN, Vriesman MH, Saps M, Rajindrajith S, Shi X, van Etten-Jamaludin FS, Di Lorenzo C, Benninga MA, Tabbers MM. Prevalence of Functional Defecation Disorders in Children: A Systematic Review and Meta-Analysis. J Pediatr. 2018 Jul;198:121-130.e6. doi: 10.1016/j.jpeds.2018.02.029. Epub 2018 Apr 12. PMID 29656863
- [Background] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632
- [Background] Tabbers MM, DiLorenzo C, Berger MY, Faure C, Langendam MW, Nurko S, Staiano A, Vandenplas Y, Benninga MA; European Society for Pediatric Gastroenterology, Hepatology, and Nutrition; North American Society for Pediatric Gastroenterology. Evaluation and treatment of functional constipation in infants and children: evidence-based recommendations from ESPGHAN and NASPGHAN. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):258-74. doi: 10.1097/MPG.0000000000000266. PMID 24345831
- [Background] Boilesen SN, Tahan S, Dias FC, Melli LCFL, de Morais MB. Water and fluid intake in the prevention and treatment of functional constipation in children and adolescents: is there evidence? J Pediatr (Rio J). 2017 Jul-Aug;93(4):320-327. doi: 10.1016/j.jped.2017.01.005. Epub 2017 Apr 25. PMID 28450053
- [Background] Santucci NR, Chogle A, Leiby A, Mascarenhas M, Borlack RE, Lee A, Perez M, Russell A, Yeh AM. Non-pharmacologic approach to pediatric constipation. Complement Ther Med. 2021 Jun;59:102711. doi: 10.1016/j.ctim.2021.102711. Epub 2021 Mar 15. PMID 33737146
- [Background] Koppen IJN, Saps M, Lavigne JV, Nurko S, Taminiau JAJM, Di Lorenzo C, Benninga MA. Recommendations for pharmacological clinical trials in children with functional constipation: The Rome foundation pediatric subcommittee on clinical trials. Neurogastroenterol Motil. 2018 Apr;30(4):e13294. doi: 10.1111/nmo.13294. Epub 2018 Jan 30. PMID 29380480